CLINICAL TRIAL: NCT01184066
Title: The ACTS Intervention to Reduce Breast Cancer Treatment Disparity
Brief Title: The Attitudes, Communication, Treatment and Support Intervention to Reduce Breast Cancer Treatment Disparity
Acronym: ACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Margaret Quinn Rosenzweig, PhD, FNP-C, AOCNP,FAAN, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 706367; RSGT-09-150-01 CPHPS (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2010-08-11; First posted 2010-08-18 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Chemotherapy; Patient Adherence; African Americans; Cancer Survivor; Decision Making; Communication; Quality of Life; Social Support; Patient Education
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance; Communication

STUDY DESIGN:
Masking Description: There was no masking. This intervention was open.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACTS Intervention (Experimental): The intervention arm are the women who received the ACTS Intervention. It is a 45 minute intervention provided by a breast cancer survivor. The intervention includes a discussion of the patient's attitudes towards chemotherapy, communication strategies with providers, the recommended treatment in accordance with tumor size and tumor characteristics
  Interventions: Behavioral: ACTS Intervention
- Usual Care (Active Comparator): This group receives care as usual.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: ACTS Intervention — ACTS (Attitudes, Communication, Treatment, Support) Intervention is a onetime intensive 45 minute intervention delivered by a black breast cancer survivor and utilizing video, graphics, teaching tools, and supportive testimony to encourage chemotherapy adherence.
  Arms: ACTS Intervention
Behavioral: Usual Care — Usual Care will consist of standard therapy education by a registered nurse in the treatment center. Education and support from clinicians are offered as needed throughout the course of cancer treatment at all participating medical oncology clinics.
  Arms: Usual Care

SUMMARY:
The ACTS (Attitudes, Communication, Treatment, Support) Intervention is a onetime, intensive psycho-educational intervention using a race-matched breast cancer survivor interventionist to: address Attitudes, including perceptions and stressors, that may impact adherence to clinical visits and treatment; encourage and model patient Communication with health care providers regarding physical and emotional needs, with attention to race-discordant situations; and provide tailored, understandable information about Treatment and its rationale. The Support component is threaded throughout the intervention via the presence of a race-matched breast cancer survivor and supportive video messages from the black community.

DETAILED DESCRIPTION:
The 5-year survival after a first diagnosis of breast cancer is 13% lower in black than in white American women, an alarming disparity that cannot be explained by stage of disease at presentation. Nonadherence to breast cancer treatment and treatment delays from diagnosis to initiation of treatment may be among the reasons for worse breast cancer outcomes in black women. This recognition is critical because it suggests that breast cancer survival disparity can be decreased through clinical interventions that increase adherence to chemotherapy. The ACTS (Attitudes, Communication, Treatment, Support) Intervention is a onetime, intensive psycho-educational intervention using a race-matched breast cancer survivor interventionist to: address Attitudes, including perceptions and stressors, that may impact adherence to clinical visits and treatment; encourage and model patient Communication with health care providers regarding physical and emotional needs, with attention to race-discordant situations; and provide tailored, understandable information about Treatment and its rationale. The Support component is threaded throughout the intervention via the presence of a race-matched breast cancer survivor and supportive video messages from the black community. This study is a randomized controlled trial that will test the efficacy of the ACTS Intervention vs. Usual Care on the primary outcomes of adherence to recommended breast cancer chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* African American, as determined by patient self report on their demographic form completed at first medical oncology visit
* Female
* Age 18 or older
* Diagnosed with invasive breast cancer
* Recommended (prescribed) chemotherapy by participating medical oncologists

Exclusion Criteria:

* Impaired cognition, as determined by a score of less than 22 on the Mini Mental Status Exam
* An inability to understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adherence to recommended breast cancer chemotherapy at the treatment midpoint. | Midpoint of the recommented chemotherapy treatment regimen.
  Midpoint chemotherapy adherence was measured by recording the chemotherapy dose received/chemotherapy dose prescribed at the treatment midpoint via medical record review for each participant in both the ACTS Intervention and Usual Care groups.
Adherence to recommended breast cancer chemotherapy at the treatment endpoint. | Endpoint of the recommented chemotherapy treatment regimen.
  Endpoint chemotherapy adherence was measured by recording the chemotherapy dose received/chemotherapy dose prescribed at the treatment endpoint via medical record review for each participant in both the ACTS Intervention and Usual Care groups.

SECONDARY OUTCOMES:
Social Support ISEL-12 | baseline (0 weeks), midpoint (6 or 12 weeks), and endpoint (12 or 24 weeks) of recommended chemotherapy regimen
  Social Support will be assessed with the Interpersonal Support Evaluation List (ISEL-12), the shortened general population form. The ISEL was designed to assess the perceived availability of four separate functions of social support as well as providing an overall support measure. The items which comprise the ISEL fall into four 10-item subscales listed as tangible, appraisal, self esteem and belonging. Scoring is based on a 5 point Likert scale test-retest data reveal correlations between .77-.86 Cronbach alpha = .86
Symptom Incidence | baseline (0 weeks), midpoint (6 or 12 weeks), and endpoint (12 or 24 weeks) of recommended chemotherapy regimen
  Symptom Occurrence and Severity Measure: The McCorkle Symptom Distress Scale (SDS) was developed in 1977 based on interviews with patients about their symptom experiences. Scores range from 1 to 5 on a Likert-type scale with 5 indicating most severe.157 Total symptom distress can be obtained as the unweighted sum of 13 items. If an item is scored as 3 or above it is considered to indicate serious distress. A cumulative score of 25 or more indicates moderate distress and any score above 33 indicates severe distress necessitating immediate intervention.149 The SDS can be administered as paper questionnaire.
Symptom Distress | baseline (0 weeks), midpoint (6 or 12 weeks), and endpoint (12 or 24 weeks) of recommended chemotherapy regimen
  Symptom Occurrence and Severity Measure: The McCorkle Symptom Distress Scale (SDS) was developed in 1977 based on interviews with patients about their symptom experiences. Scores range from 1 to 5 on a Likert-type scale with 5 indicating most severe.157 Total symptom distress can be obtained as the unweighted sum of 13 items. If an item is scored as 3 or above it is considered to indicate serious distress. A cumulative score of 25 or more indicates moderate distress and any score above 33 indicates severe distress necessitating immediate intervention.149 The SDS can be administered as paper questionnaire.
Communication of Symptoms. The Symptom Severity and Symptoms Reporting Checklist | baseline (0 weeks), midpoint (6 or 12 weeks), and endpoint (12 or 24 weeks) of recommended chemotherapy regimen
  Twenty two symptoms are assessed. If present, the patient is then asked if they reported the symptom to their doctor or nurse and if they received recommendations made by the health care team. The psychometrics for this instrument are not established. This instrument measures a key component of the ACTS Intervention, the ability to communicate distress to health care professionals. Scoring is dichotomous (yes/no) for experiencing the symptom and yes/no spoke with physician or nurse about that symptom. Total score is number of symptoms reported over number of symptoms total.
Quality of Life-FACT Functional Assessment of Cancer Therapy | baseline (0 weeks), midpoint (6 or 12 weeks), and endpoint (12 or 24 weeks) of recommended chemotherapy regimen
  The Functional Assessment of Cancer Therapy is a 27- item self-report Likert scale questionnaire comprising four subscales-physical well being, social well being, functional well-being, and emotional well-being The FACT is designed to measure health-related quality of life for individuals with cancer.147 Each item is rated from on a scale of zero to four with zero equal to "not at all" and four equal to "very much." This questionnaire requires 5-7 minutes to complete. It has been determined appropriate for use in clinical oncology settings and shown to have good validity and reliability.148 In initial psychometric evaluation, the mean score for the FACT- G was 82.05 (SD 15.86)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Q Rosenzweig, PhD,FNP-C, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - West Penn Allegheny Health System, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Overall study results will be published. Individual participant data will not be made available due to privacy issues.